CLINICAL TRIAL: NCT01880710
Title: Randomized Clinical Trial of Total Versus Subtotal Abdominal Hysterectomy
Brief Title: Total Versus Subtotal Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nykøbing Falster County Hospital (Other)
Collaborators: University of Southern Denmark (Other); Zealand University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lea Laird Andersen, MD, PhD.-student, Nykøbing Falster County Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sj-268
Record Dates: First submitted 2013-05-14; First posted 2013-06-19 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Benign Uterine Disease
Keywords: long term follow-up; urinary incontinence; pelvic organ prolapse; total versus subtotal hysterectomy
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total hysterectomy (Active Comparator): removal of the entire uterus including the cervix. open abdominal surgery. No specific procedures were asked of the surgeon. They were free to do the procedure the way they were used to doing it.
  Interventions: Procedure: Total Hysterectomy
- Subtotal Hysterectomy (Experimental): removal of the uterine body only leaving the cervix in situ. The surgeon was free to do the procedure as he was used to. The only direction was that the cervical canal should be electrocoagulated.
  Interventions: Procedure: Subtotal hysterectomy

INTERVENTIONS:
Procedure: Subtotal hysterectomy — Subtotal abdominal hysterectomy where the body of the uterus is removed but the cervix is spared.
  Arms: Subtotal Hysterectomy
Procedure: Total Hysterectomy — total abdominal hysterectomy where the body as well as the cervix of the uterus are removed.
  Arms: Total hysterectomy

SUMMARY:
319 Women undergoing hysterectomy for benign (not cancer) indications were randomly allocated to 2 types of surgery (Total (TAH) and Subtotal (SAH)) abdominal hysterectomy 15 years ago. They were followed by questionnaire at time of surgery and up to 5 years (not yet published) after the surgery and evaluated regarding following outcomes: Urinary incontinence, pain, bowel problems, per and postoperative complications, sexuality, quality of life, pelvic organ prolapse and vaginal bleeding. Now the investigators are conducting a 15 year follow up with the same out-come measures but also including physical examinations regarding Urinary incontinence, voiding difficulties, pelvic organ prolapse and problems with the cervix. The investigators' hypothesis is that several of the out-come measures will be present in more cases than earlier due to age and menopausal changes. The investigators expect more urinary incontinence in the subtotal group as this was seen at earlier follow ups. The investigators expect to find more women with pelvic organ prolapse with the physical examination than by questionnaire alone, possibly with a higher incidence in the subtotal group.

DETAILED DESCRIPTION:
The study included women who were offered a hysterectomy for benign uterine disease such as: metrorrhagia, menorrhagia, fibroids, endometriosis,and pelvic pain. Women in need of hysterectomy for malignant disease or because of prolapse of the uterus were not included. They were followed up by a questionnaire covering all outcome measures as described above. Background information was registered in a second questionnaire prior to surgery. All gynaecological departments in Denmark were invited to join the trial. 11 departments contributed randomized patients to the trial.

the results up to 1 year after surgery have been published, links can be found in the citation list. The results from the 5 year follow up have not yet been published.

The questionnaire used in this trial consists of the validated SF-36 (Short Form 36) quality of life questionnaire as well as a thorough questionnaire regarding the outcome measures described elsewhere. The entire questionnaire was validated prior to the beginning of the trial.

A second questionnaire has been added in the 15 year follow up: PFDI-20(Pelvic Floor Distress Inventory 20). The investigators included this, as it is more thorough regarding pelvic organ prolapse and in particular a "bother" measure than the original questionnaire.

The 20 min. pad-weighing test has been tested against the 1 hour gold-standard used by the ICS (International Continence Society) and has been found to give comparable results.

ELIGIBILITY:
Inclusion Criteria:

-Women undergoing abdominal hysterectomy for benign uterine disease at a gynaecological department in Denmark (15 years ago)

Exclusion Criteria:

* malignant disease
* mental disease
* diabetes
* neurological disease
* not able to read and write Danish
* pelvic organ prolapse as the reason for hysterectomy
* prior surgery for urinary incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change in Urinary incontinence from baseline (preoperatively) | 2 months, 6months, 1, 5 and 15 years postoperatively
  urinary incontinence measured by questionnaire filled out by the participants at each time point as well as a more objective measure: pad weighing test and voiding diary at 15 years

SECONDARY OUTCOMES:
pelvic organ prolapse | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  subjective measure by questionnaire at each time point as well as objective measure by POP-Q measurement at 15 years
cervical problems in the SAH group | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  questionnaire regarding bleeding at each time point, pap-smear regarding dysplasia at 15 years discharge summaries from hospital admissions/contacts regarding cervical problems.
voiding difficulties and LUTS (Lower Urinary Tract Symptoms) | preoperatively, 2 months, 6 months, 1, 5 and 15 years postoperatively
  covered by the questionnaire at each time point regarding urinary tract infections and problems emptying the bladder. In addition the 15 year follow up consists of uroflow, dip-stick for urinary infection as well as post-voiding ultrasound of the bladder to detect urinary retention.

OTHER OUTCOMES:
quality of life | preoperatively, 2 months, 6months, 1 and 15 years postoperatively
  SF-36 questionnaire at each time point
sexuality | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  questionnaire at each time point
pelvic pain | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  questionnaire at each time point
bowel problems | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  questionnaire at each time point
per- and postoperative complications | preoperatively, 2 months, 6months, 1, 5 and 15 years postoperatively
  questionnaire at each time points and case records regarding related surgery (hernia, bowel obstruction, removal of the cervix, surgery for urinary incontinence and pelvic organ prolapse)looked up in the clinical registry

CONTACTS AND LOCATIONS:
Overall Officials: Lea L Andersen, MD, Principal Investigator — Nykoebing Falster County Hospital; Helga ME Gimbel, Dr.med.sci., Study Director — University of Southern Denmark
Locations (1):
- Nykoebing Falster County Hospital, Nykoebing Falster, Region Sjælland, Denmark

REFERENCES:
- [Background] Gimbel H, Zobbe V, Ottesen BS, Tabor A. Randomized clinical trial of total vs. subtotal hysterectomy: validity of the trial questionnaire. Acta Obstet Gynecol Scand. 2002 Oct;81(10):968-74. doi: 10.1034/j.1600-0412.2002.811012.x. PMID 12366489
- [Result] Gimbel H, Zobbe V, Andersen BJ, Sorensen HC, Toftager-Larsen K, Sidenius K, Moller N, Madsen EM, Vejtorp M, Clausen H, Rosgaard A, Villumsen J, Gluud C, Ottesen BS, Tabor A. Lower urinary tract symptoms after total and subtotal hysterectomy: results of a randomized controlled trial. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Jul-Aug;16(4):257-62. doi: 10.1007/s00192-005-1291-8. PMID 16220584
- [Result] Gimbel H, Zobbe V, Andersen BM, Filtenborg T, Gluud C, Tabor A. Randomised controlled trial of total compared with subtotal hysterectomy with one-year follow up results. BJOG. 2003 Dec;110(12):1088-98. PMID 14664880
- [Result] Zobbe V, Gimbel H, Andersen BM, Filtenborg T, Jakobsen K, Sorensen HC, Toftager-Larsen K, Sidenius K, Moller N, Madsen EM, Vejtorp M, Clausen H, Rosgaard A, Gluud C, Ottesen BS, Tabor A. Sexuality after total vs. subtotal hysterectomy. Acta Obstet Gynecol Scand. 2004 Feb;83(2):191-6. doi: 10.1111/j.0001-6349.2004.00311.x. PMID 14756739
- [Derived] Andersen LL, Moller LM, Gimbel HM. Low adherence to cervical cancer screening after subtotal hysterectomy. Dan Med J. 2015 Dec;62(12):A5165. PMID 26621394
- [Derived] Andersen LL, Alling Moller LM, Gimbel HM. Objective comparison of subtotal vs. total abdominal hysterectomy regarding pelvic organ prolapse and urinary incontinence: a randomized controlled trial with 14-year follow-up. Eur J Obstet Gynecol Reprod Biol. 2015 Oct;193:40-5. doi: 10.1016/j.ejogrb.2015.06.033. Epub 2015 Jul 9. PMID 26231437
- [Derived] Andersen LL, Moller LM, Gimbel H; Danish Hysterectomy Trial Group. Lower urinary tract symptoms after subtotal versus total abdominal hysterectomy: exploratory analyses from a randomized clinical trial with a 14-year follow-up. Int Urogynecol J. 2015 Dec;26(12):1767-72. doi: 10.1007/s00192-015-2778-6. Epub 2015 Jul 28. PMID 26215904
- [Derived] Andersen LL, Zobbe V, Ottesen B, Gluud C, Tabor A, Gimbel H; Danish Hysterectomy Trial Group. Five-year follow up of a randomised controlled trial comparing subtotal with total abdominal hysterectomy. BJOG. 2015 May;122(6):851-857. doi: 10.1111/1471-0528.12914. Epub 2014 Jun 11. PMID 24917531